CLINICAL TRIAL: NCT00769938
Title: What is the Optimal antiplatElet & Anticoagulant Therapy in Patients With Oral Anticoagulation and Coronary StenTing
Brief Title: WOEST ( What is the Optimal antiplatElet & Anticoagulant Therapy in Patients With Oral Anticoagulation and Coronary StenTing)
Acronym: WOEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Responsible Party: Principal Investigator, W. Dewilde, Dr, R&D Cardiologie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDC-2008-03
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Anticoagulants; Platelet Aggregation Inhibitors; Stents; Atrial Fibrillation
Keywords: Atrial fibrillation; Percutaneous coronary stenting; Bleeding complications; Triple therapy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin + clopidogrel + oral anticoagulation (Active Comparator)
  Interventions: Device: PCI (percutaneous coronary intervention)
- Oral anticoagulants + clopidogrel (Active Comparator)
  Interventions: Device: PCI (percutaneous coronary intervention)

INTERVENTIONS:
Device: PCI (percutaneous coronary intervention) — only patients scheduled for PCI can be included tough this intervention would also take place without this study. What we want to study is the difference in outcome after a little change in the antithrombotic treatment

SUMMARY:
The study will assess the hypothesis that the combination warfarin & clopidogrel 75 mg/day is superior to triple therapy (warfarin + clopidogrel 75mg/day + aspirin 80mg/day) with respect to bleeding complications while equally safe with respect to the prevention of thrombotic complications in patients with both indications for warfarin use and dual antiplatelet (clopidogrel 75mg/day + aspirin 80mg/day) treatment.

DETAILED DESCRIPTION:
Chronic oral antithrombotic treatment is necessary in patients with mechanical heart valves and in the majority of patients with atrial fibrillation. When these patients have to undergo Percutaneous Coronary Intervention (PCI) with stenting, there is also an indication for treatment with aspirin and clopidogrel. However, triple therapy is known to augment the risk for bleeding complications.Unfortunately, no prospective data are available to solve this issue. Nevertheless, it all comes down to finding the ideal therapy in patients with both atrial fibrillation and percutaneous intervention to prevent thrombotic complications (e.g. stent thrombosis) without increasing the risk of bleeding. This prospective randomised study will assess the hypothesis that in patients on warfarin therapy and indication for elective percutaneous intervention, the combination warfarin & clopidogrel 75 mg/day is superior to triple therapy treatment in reducing the risk of bleeds while equally safe with respect to the prevention of thrombotic complications

ELIGIBILITY:
Inclusion Criteria:

* Patients is on oral anticoagulation therapy and this will be continued throughout the period of 1 year-and deployment of at least 1 coronary stent (bare metal stent (BMS) or drug eluting stent (DES)). -age of more than 18 years

Exclusion Criteria:

* cardiogenic shock,
* contra-indication for aspirin or clopidogrel
* allergy to aspirin or clopidogrel,
* documented peptic ulcer disease within the previous six months,
* pregnancy and
* previous intracerebral haemorrhage or
* significant thrombocytopenia (platelet count < 50x10 9/L).
* major bleeding according to timi criteria within the past 12 months
* age > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2008-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The combined end point of minor, moderate or major bleeding complications during the initial hospitalization & one year follow-up. (TIMI & GUSTO criteria). | 1 year

SECONDARY OUTCOMES:
The combined event of death, myocardial infarction, stroke, systemic embolization & target vessel revascularisation and the individual components of the composite primary and secondary endpoints. | 1 year

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (5):
  - UZ KU Leuven, Leuven, Leuven
  - OLV Aalst, Aalst
  - UZ Antwerpen, Antwerp
  - ZOL, Genk
  - Maria Middelares, Ghent
- Netherlands (10):
  - MCA Alkmaar, Alkmaar
  - Academisch Medisch Centrum Amsterdam, Amsterdam
  - OLVG, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina Ziekenhuis, Eindhoven
  - UMCG, Groningen
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Zuiderziekenhuis, Rotterdam
  - Twee Steden Ziekenhuis, Tlibrug
  - Isala klinieken, Zwolle

REFERENCES:
- [Derived] Dewilde WJ, Janssen PW, Kelder JC, Verheugt FW, De Smet BJ, Adriaenssens T, Vrolix M, Brueren GB, Van Mieghem C, Cornelis K, Vos J, Breet NJ, ten Berg JM. Uninterrupted oral anticoagulation versus bridging in patients with long-term oral anticoagulation during percutaneous coronary intervention: subgroup analysis from the WOEST trial. EuroIntervention. 2015 Aug;11(4):381-90. doi: 10.4244/EIJY14M06_07. PMID 24970794
- [Derived] Dewilde WJ, Oirbans T, Verheugt FW, Kelder JC, De Smet BJ, Herrman JP, Adriaenssens T, Vrolix M, Heestermans AA, Vis MM, Tijsen JG, van 't Hof AW, ten Berg JM; WOEST study investigators. Use of clopidogrel with or without aspirin in patients taking oral anticoagulant therapy and undergoing percutaneous coronary intervention: an open-label, randomised, controlled trial. Lancet. 2013 Mar 30;381(9872):1107-15. doi: 10.1016/S0140-6736(12)62177-1. Epub 2013 Feb 13. PMID 23415013
- [Derived] Dewilde W, Berg JT. Design and rationale of the WOEST trial: What is the Optimal antiplatElet and anticoagulant therapy in patients with oral anticoagulation and coronary StenTing (WOEST). Am Heart J. 2009 Nov;158(5):713-8. doi: 10.1016/j.ahj.2009.09.001. PMID 19853687